CLINICAL TRIAL: NCT04069507
Title: Healthy Hip Study: Predictors of Successful Conservative Management for Pre-arthritic Hip Disorders: Prospective Study
Brief Title: Healthy Hip Study: Conservative Management for Pre-arthritic Hip Disorders
Acronym: HHS
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Abby Cheng, Assistant Professor, Washington University School of Medicine
Other Study IDs: 201807150; 1K23AR074520-01A1 (NIH)
Record Dates: First submitted 2019-08-21; First posted 2019-08-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Femoroacetabular Impingement; Acetabular Dysplasia; Acetabular Labrum Tear; Hip Pain; Rehabilitation
Keywords: Biopsychosocial health; Clinical prediction tool; Patient-reported outcomes; Movement pattern training
MeSH Terms: conditions — Femoracetabular Impingement; Hip Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Pre-arthritic hip disorders can cause pain, interfere with daily activities and exercise, and lead to the development of osteoarthritis in young adults. Surgical and conservative treatment options are being developed and studied, but it is currently unclear why some patients improve with a particular treatment plan while others do not. The goal of this research project is to develop a tool that predicts which combination of treatment options will be most effective for each individual patient.

DETAILED DESCRIPTION:
Significance: Pre-arthritic hip disorders (PAHD) are bony and soft tissue hip morphologies that predispose adolescents and young adults to developing hip pain, chronic impairment, and early osteoarthritis (OA). Proper management may prevent these sequelae, but current evidence, especially regarding non-operative treatment options, is limited.

Innovation: The majority of PAHD has so far addressed identification and correction of abnormal hip anatomy via surgical management. However, a growing body of evidence suggests that several other variables including patients' functional goals, movement patterns, and psychological profiles also affect their symptomatology. These risk factors are modifiable but are not routinely or adequately addressed. The innovation of this project is to improve patient outcomes by evaluating patients with a more comprehensive, patient-specific approach than is currently the standard of care.

Purpose: The purpose of this project is to identify predictors of response to non-operative PAHD treatment options and to synthesize these predictors into a clinical prediction tool that informs non-operative one-year outcomes using data available during patients' initial evaluation. In this prospective observational study, patients who present to an orthopedic physician for PAHD will be provided instruction on movement pattern training, which is a standardized activity modification protocol that addresses how patients perform routine and strenuous activities in order to reduce hip pain. It has proven to be efficacious in a randomized trial setting, but it is not yet widely discussed by physicians in the clinic setting. Patients will report adherence and response to the movement pattern training at scheduled intervals for 12 weeks, and they will also report persistent hip-related dysfunction and/or progression to surgery at 6 and 12 months. A clinical prediction tool of one-year outcomes will be developed using patients' demographics, biopsychosocial profile, movement and activity patterns, and anatomy as candidate predictors. The analysis will also determine a minimum combination of patient-reported outcome measures (PROMs) that reduces survey burden while maintaining similar predictive utility when compared to administration of a full battery of hip-specific and general health PROMs.

Impact: This study is the first step in creating and validating a clinical prediction tool which will guide management for patients with pre-arthritic hip disorders. This line of research will equip clinicians to provide more accurate prognostic counseling at initial evaluation so that an informed shared decision can be made with the patient and initiation of an appropriate comprehensive management plan can be expedited.

ELIGIBILITY:
Inclusion Criteria:

* Clinically suspected intra-articular hip joint pain
* One or more of the following radiographic/MRI findings: Femoroacetabular impingement, acetabular dysplasia, acetabular labral tear, acetabular retroversion, femoral anteversion, hip microinstability, and/or normal radiographs

Exclusion Criteria:

* Surgery recommended and/or scheduled at initial clinic evaluation
* "At-risk" acetabular dysplasia (Lateral center edge angle < 15 degrees)
* Other intra-articular hip diagnoses including: Slipped capital femoral epiphysis, Legg-Calve-Perthes disease, Avascular necrosis
* Moderate or severe hip osteoarthritis (Tonnis grade 2 or 3)
* Hip/pelvis weakness from brain/nerve disorder (Ex: lumbosacral radiculopathy with weakness, cerebral palsy)
* Previous same-side hip surgery, hip fracture, hip infection, and/or hip tumor
* Inflammatory arthropathy
* Known pregnancy

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be recruited from patients who present to a single tertiary care academic orthopedic department. Potentially eligible patients will have presented to an orthopedic surgeon or sports medicine physiatrist for a new evaluation of hip pain.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2024-09-22 (Actual)

PRIMARY OUTCOMES:
Rate of successful conservative management | 1 Year
  Percentage of participants who self-report satisfactory overall hip symptoms and no plan to proceed with surgery. The rate will be adjusted for patients' baseline demographics, severity of hip symptoms, biopsychosocial profile, hypermobility profile, movement and activity patterns, and hip anatomy.

SECONDARY OUTCOMES:
Rate of adherence and symptom response to movement pattern training | 12 Weeks
  Percentage of participants who are adherent to the movement pattern training protocol for at least one study interval and who report at least moderate symptomatic improvement on a Global Rating of Change scale as a result of adherence
Rate of clinically meaningful improvement with conservative management | 1 Year
  Percentage of participants who do not proceed to hip surgery and who either self-report satisfactory overall hip symptoms or meet the minimal clinically important difference (MCID) on the International Hip Outcome Tool-12 (iHOT-12)

CONTACTS AND LOCATIONS:
Overall Officials: Abby L Cheng, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators are amenable to sharing individual participant data (IPD) when all anticipated data analyses are complete. However, the data generated from this study may be used for future validation efforts of new versions of the clinical prediction tool. The IPD will likely not be made available until there is reasonable confidence that no further data analyses are planned.

REFERENCES:
- [Background] Harris-Hayes M, Czuppon S, Van Dillen LR, Steger-May K, Sahrmann S, Schootman M, Salsich GB, Clohisy JC, Mueller MJ. Movement-Pattern Training to Improve Function in People With Chronic Hip Joint Pain: A Feasibility Randomized Clinical Trial. J Orthop Sports Phys Ther. 2016 Jun;46(6):452-61. doi: 10.2519/jospt.2016.6279. Epub 2016 Apr 26. PMID 27117727
- [Background] Prather H, Creighton A, Sorenson C, Simpson S, Reese M, Hunt D, Rho M. Anxiety and Insomnia in Young and Middle-Aged Adult Hip Pain Patients With and Without Femoroacetabular Impingement and Developmental Hip Dysplasia. PM R. 2018 May;10(5):455-461. doi: 10.1016/j.pmrj.2017.10.007. Epub 2017 Oct 27. PMID 29111466
- [Background] Hunt D, Prather H, Harris Hayes M, Clohisy JC. Clinical outcomes analysis of conservative and surgical treatment of patients with clinical indications of prearthritic, intra-articular hip disorders. PM R. 2012 Jul;4(7):479-87. doi: 10.1016/j.pmrj.2012.03.012. Epub 2012 May 16. PMID 22595328
- [Background] Prather H, Decker G, Bonnette M, Simpson S, Hunt D, Sahrmann S, Cheng A, Nepple J. Hip Radiograph Findings in Patients Aged 40 Years and Under with Posterior Pelvic Pain. PM R. 2019 Aug;11 Suppl 1:S46-S53. doi: 10.1002/pmrj.12180. Epub 2019 Jul 25. PMID 31059595
- [Background] Prather H, Cheng A, Steger-May K, Maheshwari V, VanDillen L. Association of Hip Radiograph Findings With Pain and Function in Patients Presenting With Low Back Pain. PM R. 2018 Jan;10(1):11-18. doi: 10.1016/j.pmrj.2017.06.003. Epub 2017 Jun 16. PMID 28629805
- [Background] Prather H, Cheng A, Steger-May K, Maheshwari V, Van Dillen L. Hip and Lumbar Spine Physical Examination Findings in People Presenting With Low Back Pain, With or Without Lower Extremity Pain. J Orthop Sports Phys Ther. 2017 Mar;47(3):163-172. doi: 10.2519/jospt.2017.6567. Epub 2017 Feb 3. PMID 28158964
- [Derived] Cheng AL, Pashos MM, Hannemann AJ, Brady BK, Huecker JB, Steger-May K, Prather H, Clohisy JC, Harris-Hayes M. Predictors and rate of satisfactory response to nonoperative management for nonarthritic hip-related pain. PM R. 2026 Jan 27. doi: 10.1002/pmrj.70085. Online ahead of print. PMID 41589432